CLINICAL TRIAL: NCT06335446
Title: Identification, Electro-mechanical Characterisation and Ablation of Driver Regions in Persistent Atrial Fibrillation (STAR Mapping)
Brief Title: Identification, Electro-mechanical Characterisation and Ablation of Driver Regions in Persistent Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 011040- AT validation phase; PG/16/10/32016 (Other Grant/Funding Number: British Heart Foundation)
Record Dates: First submitted 2018-01-17; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Atrial Tachycardia
Keywords: Atrial tachycardia, Electrogram, Ablation, Drivers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Atrial tachycardia- validation phase: The group will consist of patients with AT (whether de novo or occurring post AF ablation) that are undergoing catheter ablation.
  Interventions: Other: Novel mapping algorithm

INTERVENTIONS:
Other: Novel mapping algorithm — Signals will be collected during the catheter ablation. These signals STAR maps will be created post procedure and these will be compared to the conventional maps used during the atrial tachycardia ablation. This will be used to validate the STAR maps created.
  Other Names: STAR MAPPING

SUMMARY:
Atrial fibrillation (AF) is the most common sustained heart rhythm abnormality. Its incidence is increasing partly due to the aging population and it has been referred to as a growing epidemic. AF results in irregular contractions of the heart causing unpleasant symptoms of palpitations and increasing the risk of stroke, heart failure and death. Percutaneous catheter ablation is a safe treatment option in symptomatic patients with AF. The success rate of these procedures have improved with time due to our better understanding of AF, development of new techniques and technology, and greater physician experience. However, the success rate of these procedures still only remains around 70%. This is secondary to our limited ability to find the areas that drive AF.

STAR mapping is a novel mapping system that has been developed with a view of better identifying the sites that drive AF through taking into account the mechanisms of AF we have so far demonstrated. To validate this mapping system we aim to use it in patients with atrial tachycardia (AT), which is a heart rhythm abnormality of which the mechanism can be readily identified with the existing mapping systems used in clinical practice. We will demonstrate that the STAR mapping algorithm can effectively map AT.

DETAILED DESCRIPTION:
AT is a heart rhythm that currently can be effectively mapped and ablated using existing mapping systems. The mechanism of this heart rhythm is well understood.

Patients that are scheduled for a catheter ablation for AT by their Electrophysiologist will be enrolled into the study. The patient will have the procedure under local anaesthetics/sedation or general anaesthetic depending on their clinical need.

During the procedure tubes will be passed into the left upper chamber of the heart through the groin. Through these tubes catheters will be used to create a geometry of the heart chamber. Following this, in half of the patients a basket catheter with 64 electrodes will be positioned in the upper chamber whilst conventional catheters will be used in the other half of the patients. The aim of this is to demonstrate that the STAR mapping can be used with multiple mapping catheters. Signals i.e. electrograms will then be collected and used with the STAR mapping algorithm. The AT will then be effectively mapped and ablated with a conventional mapping system. The STAR mapping will then be used for post processing after the case to map the AT and will be compared to the maps generated by the conventional system. This will enable validation of the STAR mapping system.

ELIGIBILITY:
Inclusion Criteria:

1. Patients able to provide informed consent
2. Patients with AT (whether de novo or occurring post AF ablation)

Exclusion Criteria:

1. Unwillingness to sign consent
2. Age <18 years old
3. Contraindications for catheter ablation procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AT (whether de novo or occurring post AF ablation) undergoing catheter ablation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-10; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
STAR maps compared to conventional maps | At procedure
  The STAR maps demonstrating the source of the AT correlate with the maps created by the conventional mapping system.

CONTACTS AND LOCATIONS:
Locations (1):
- Barts Heart Centre, London, United Kingdom